CLINICAL TRIAL: NCT00590954
Title: Clinical and Molecular-Metabolic Phase II Trial of Perifosine for Recurrent/Progressive Malignant Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Keryx Biopharmaceuticals (Industry); Keryx / AOI Pharmaceuticals, Inc. (Industry); Online Collaborative Oncology Group (Other); University of Wisconsin, Madison (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-044; NCT00400920 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-11

CONDITIONS: Malignant Gliomas; CNS; Brain Cancer; Cancer
Keywords: Malignant Gliomas; CNS; Brain Cancer; Cancer; Perifosine
MeSH Terms: conditions — Glioma; Brain Neoplasms; Neoplasms | interventions — perifosine; octadecyl-(N,N-dimethylpiperidino-4-yl)-phosphate

ARMS (1):
- Treatment (Experimental): Following a diagnosis of tumor recurrence or progression, all patients will receive perifosine monotherapy until toxicity, progression, or death.
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — Dosing will be continuous, and for the purpose of this trial a cycle will be defined as 28 days. Perifosine will be given as a 600 mg loading dose on day 1. The loading dose will be divided into 4 equal doses of 150 mg each. The first 3 doses should be given with food in the adult day hospital to allow intravenous antiemetic prophylaxis, and 4th dose at bedtime at home. The interval between doses of perifosine should be no less than 4 hours. On day 2, patients will start the maintenance dose of 100 mg daily at bedtime at home.
  In addition to baseline serum, all patients will have weekly serum drawn during weeks 2-4.
  Other Names: NSC 639966, D21266, KRX-0401

SUMMARY:
The purpose of this study is to test the effectiveness of perifosine in preventing further tumor growth using the established optimal dose of the drug. A second goal is to determine if perifosine can block the molecules in the tumor that drive it to divide and grow.

DETAILED DESCRIPTION:
This is a phase II study of the small molecule inhibitor perifosine (NSC 639966, D21266, KRX-0401) in the treatment of patients with recurrent glioblastoma multiforme (GBM) and other recurrent malignant gliomas. The goal of the phase II study is to determine efficacy as measured by the progressionfree survival rate after 6 months of treatment. Secondary goals include determination of molecular and metabolic effects of perifosine by tissue analysis and PET imaging.

In addition, when cytoreductive surgery is recommended as part of the standard of care at study entry, patients will be considered for a "surgical arm." In this case, patients will receive perifosine for 5-10 days before surgery during which tumor will be aliquoted both for diagnostic purposes and for molecular effects of the drug in vivo and for analysis of drug penetration into tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have shown unequivocal evidence for tumor progression by MRI or CT scan.
* Patients must be on a stable or decreasing dose of corticosteroids for a minimum of 5 days before the baseline MRI and PET scans.
* Patients must have failed prior radiation therapy.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery (including gamma-knife or cyber-knife) must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, and/or MR spectroscopy, and/or MR Perfusion, and/or surgical documentation of disease.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
* Age > 18 years old, and with a life expectancy > 8 weeks.
* Karnofsky Performance Status ≥ 50%
* Patients must have recovered from all acute toxicities from prior therapies. At least 28 days must have elapsed since prior radiation.
* Patients must have adequate bone marrow function
* Patients must agree to practice adequate contraception.

Exclusion Criteria:

* Patients must not be taking EIAEDs
* Patients must not have any significant medical illnesses or other history that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have active infection or serious intercurrent medical illness.
* HIV-Positive patients receiving combination anti-retroviral therapy are excluded from the study due to possible retro-viral drug interactions.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Following a diagnosis of tumor recurrence or progression, all patients will receive perifosine monotherapy until toxicity, progression, or death.
  Perifosine: Dosing will be continuous, and for the purpose of this trial a cycle will be defined as 28 days. Perifosine will be given as a 600 mg loading dose on day 1. The loading dose will be divided into 4 equal doses of 150 mg each. The first 3 doses should be given with food in the adult day hospital to allow intravenous antiemetic prophylaxis, and 4th dose at bedtime at home. The interval between doses of perifosine should be no less than 4 hours. On day 2, patients will start the maintenance dose of 100 mg daily at bedtime at home.
  In addition to baseline serum, all patients will have weekly serum drawn during weeks 2-4.
Period: Overall Study
Arm/Group | Treatment
Started | 32
Completed | 30
Not Completed | 2
Not completed — Inevaluable | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 51 [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Determine the Efficacy of Perifosine in Patients With Recurrent/Progressive GBMs Not Taking EIAEDs as Measured by 6 Month Progression Free Survival/PFS.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Glioblastoma; Anaplastic Glioma: Following a diagnosis of tumor recurrence or progression, all patients will receive perifosine monotherapy until toxicity, progression, or death.
  Perifosine: Dosing will be continuous, and for the purpose of this trial a cycle will be defined as 28 days. Perifosine will be given as a 600 mg loading dose on day 1. The loading dose will be divided into 4 equal doses of 150 mg each. The first 3 doses should be given with food in the adult day hospital to allow intravenous antiemetic prophylaxis, and 4th dose at bedtime at home. The interval between doses of perifosine should be no less than 4 hours. On day 2, patients will start the maintenance dose of 100 mg daily at bedtime at home.
  In addition to baseline serum, all patients will have weekly serum drawn during weeks 2-4.
Arm/Group | Glioblastoma | Anaplastic Glioma
Number analyzed (Participants) | 16 | 14
months | 1.58 [1.08 to 1.84] | 2.12 [1.84 to 12.79]

2. Secondary Outcome: Determine Metabolic Effects of Perifosine on Malignant Gliomas by PET Imaging
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 30/32
Serious Adverse Events (participants affected / at risk) | 22/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=32)
Confusion (Psychiatric disorders) | 2
Death not assoc w CTCAE term- Death NOS (General disorders) | 1
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 1
Hemorrhage, CNS (Nervous system disorders) | 1
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 1
Infection w/ Gr 3/4 neut, Wound (Infections and infestations) | 1
Memory impairment (Nervous system disorders) | 1
Mood alteration - Agitation (Psychiatric disorders) | 1
Muscle weakness - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness - Left-sided (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness - Whole body/general (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Neurology - Other (specify) (Nervous system disorders) | 3
Nrpthy:cranl-CN X Mtr-palate;phrynx,lrynx (Nervous system disorders) | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain - Pain NOS (General disorders) | 1
Pain - Stomach (Gastrointestinal disorders) | 1
Platelets (Investigations) | 1
Secondary malig-poss related to ca txt specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Seizure (Nervous system disorders) | 13
Somnolence/dprssd level of conscious (Nervous system disorders) | 3
Speech impairment (Nervous system disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=32)
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Lymphopenia (Investigations) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Increased alanine aminotransferase (Investigations) | 13
Fatigue (General disorders) | 10
Thrombocytopenia (Investigations) | 9
Diarrhea (Gastrointestinal disorders) | 7
Elevated aspartate transaminase (AST) (Investigations) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Leukopenia (Investigations) | 5
Nausea (Gastrointestinal disorders) | 5
Alkaline phosphatase (Investigations) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT00590954/Prot_SAP_000.pdf